CLINICAL TRIAL: NCT03826745
Title: The CHYMASE Angiotensin-(1-12) Axis in Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trinity Hypertension & Metabolic Research Institute (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Principal Investigator, Henry Anthony Punzi, Medical Director, Trinity Hypertension & Metabolic Research Institute
Other Study IDs: PMC-60-009
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Plasma and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Plasma/Urine — Plasma of normal male and female normotensive, hypertensive, and/or resistant hypertensive subjects.

SUMMARY:
Study is to evaluate the Chymase Angiotensin-(1-12) in cardiovascular disease

DETAILED DESCRIPTION:
Study is to determine the presence of the human sequence on Ang-(1-12) in the plasma of normal male and female normotensive, hypertensive and/or resistant hypertensive subjects.

To measure concentrations of Ang-(1-12) in either serum or spot urine collections from male and female normal, hypertensive and/or resistant hypertensive subjects.

To assess whether chymase activity can be detected in human serum and urine using the radiolabeled amino acid sequence of 1251-Ang-(1-12)

ELIGIBILITY:
Inclusion Criteria:

* Cable of reading, comprehending the consent process and providing written informed consent to participate in the study.
* Male or female equal/over 40 years of age.
* Currently being treated with 3 medications and are not at goal seated, Blood pressure of Systolic blood pressure less 140 mmHg and/or Diastolic blood pressure less 90 mmHg (Diabetic patients goal seated blood pressure- Systolic blood pressure less 130 and/or Diastolic blood pressure less 80) OR
* Stage I-II hypertension defined as a baseline mean seated cuff Diastolic blood pressure of equal/over 90 mmHg and equal/less 115 mmHg and/or Systolic blood pressure equal/over 140 mmHg and equal/less 180 mmHg OR
* Normotensive patients defined as a blood pressure less 140/90 mmHg
* Women may be enrolled if all three of the following criteria are met:
* Have a negative urine pregnancy test at screening, for females of childbearing potential
* Are not breastfeeding
* Do not plan t become pregnant during the study
* And if one of the following three criteria is met:
* Have had a hysterectomy or tubal ligation at least 6 months prior to signing the informed consent form
* Have been postmenopausal for at least 1 year
* Are of childbearing potential and will practice one of the following methods of birth control throughout the study: oral, patch, injectable, or implantable hormone contraception, intrauterine device, diaphragm plus spermicide or female condom plus spermicide. Abstinence, partner's vasectomy are not acceptable methods of contraception.

Exclusion Criteria:

* Patients with severe hypertension (mean seated cuff Diastolic blood pressure over 115 mmHg or mean seated Systolic blood pressure over 180 mmHg) or any form of secondary hypertension at time of screening.
* Patients within the past 6 months with a history of hypertensive encephalopathy, stroke or transient ischemic attack.
* Patients within the last 6 months with a history of myocardial infarction, percutaneous transluminal coronary revascularization, coronary bypass graft, valvular surgery or unstable angina.
* Patients with a history of heart block greater than First Degree Sino atrial Block, Wolff-Parkinson-White Syndrome, Sick Sinus Syndrome, Atrial Fibrillation, Atrial Flutter, Congestive Heart Failure, or other manifestations of clinically significant cardiac valvular disease.
* Patients with hemodynamically significant cardiac valvular disease.
* Patients with evidence of significant chronic renal impairment as indicated by a serum creatinine of over 2.5mmg/dl at Visit 1.
* Patients with evidence of liver disease as indicated by Aspartate transaminase (Serum glutamic oxaloacetic) or Alanine aminotransferase (Serum glutamic pyruvic transaminase) over 2.5 times or total bilirubin over 1.5 times, the upper limit of the laboratory normal range at Visit 1.
* Patients who demonstrate other laboratory test values deviating from the normal range which are considered to be clinically significant by the investigator.
* Patients with insulin and non-insulin dependent diabetes mellitus not controlled on diet, insulin or oral hypoglycemic as defined by a Hemoglobin A1c over 10.5 % at Visit 1.
* Severe psychological or emotional condition which may interfere with participation in the study.
* History of or current use of illicit drugs or alcohol abuse.
* Participation in a clinical trial and taking any investigational drug within 30 days prior to enrolling into the study (Visit 1).
* A physical condition that would limit accurate Blood pressure measurement.
* Any other medical condition which, in the Investigator's opinion, may render the patient unable to complete the study or which would interfere with optimal participation in the study or produce significant risk to the patient.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 normotensive subjects (40-50% females) aged 40 years and above, 25 untreated or treated essential hypertensive subject (40-50%) females) age 40 years and above, and 25 subjects with diagnosis of resistant hypertension (blood pressure not controlled on 3 or more drugs) (40-50% female) aged 40 years and above.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of Ang-(1-12) in Human Plasma/Urine | one day
  Determine the presence of the human sequence of Ang-(1-12) in the plasma of normal male and female normotensive, hypertensive and/or resistant hypertensive subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Henry A Punzi, MD, Principal Investigator — Punzi Medical Center
Locations (1):
- Punzi Medical Center, Carrollton, Texas, United States

IPD SHARING:
Plan to Share IPD: No